CLINICAL TRIAL: NCT02621892
Title: A 12-Week, Randomized, Double-Blind, Placebo-Controlled Study With a 4-Week Randomized Withdrawal Period to Evaluate the Efficacy and Safety of Tenapanor for the Treatment of Constipation-Predominant Irritable Bowel Syndrome (IBS-C)
Brief Title: A 12-Week Study With a 4-Week Randomized Withdrawal Period to Evaluate the Efficacy and Safety of Tenapanor for the Treatment of IBS-C
Acronym: T3MPO-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TEN-01-301
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Constipation Predominant Irritable Bowel Syndrome
MeSH Terms: interventions — tenapanor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 50mg BID (Experimental): Tenapanor
  Interventions: Drug: Tenapanor
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tenapanor
  Other Names: RDX5791; AZD1722
  Arms: 50mg BID
Drug: Placebo
  Arms: Placebo

SUMMARY:
This phase 3, 12-week, randomized, double-blind, placebo-controlled, multi-center study will evaluate the safety and efficacy of tenapanor in subjects with constipation-predominant irritable bowel syndrome (IBS-C) as defined by the ROME III criteria and who have active disease as determined after a two-week screening period. Subjects who qualify and are randomized into the study will either receive 50mg BID of tenapanor or placebo BID for 12 week treatment period and then undergo a 4 week placebo controlled randomized withdrawal.

DETAILED DESCRIPTION:
During the 12-week treatment period, subjects will record daily assessments including: frequency and timing of bowel movements; sensation and complete bowel emptying; consistency of bowel movements; degree of straining, worst abdominal pain, abdominal discomfort, abdominal bloating, abdominal fullness and abdominal cramping. Subjects will also record weekly assessments including: adequate relief of IBS severity, and constipation severity.

At the end of the 12-week treatment period, there will be a 4-week randomized withdrawal period in which subjects who complete the study in Tenapanor group will be randomized to either Tenapanor 50mg BID or placebo BID (1:1) and subjects who complete the study in the placebo group will be assigned to receive Tenapanor 50mg BID.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old
* Females must be of non-childbearing potential; If of child-bearing potential, must have negative pregnancy test and confirm the use of one of the appropriate means of contraception.
* Males must agree to use an appropriate method of barrier contraception or have documented surgical sterilization
* Subject meets definition of IBS-C using Rome III Criteria for the Diagnosis of IBS
* A colonoscopy based on AGA guidelines; every 10 years at ≥ 50 years old, or the occurrence of any warning signs

Exclusion Criteria:

* Functional diarrhea as defined by Rome III criteria
* IBS with diarrhea (IBS-D), mixed IBS (IBS-M), or unsubtyped IBS as defined by Rome III criteria
* Diagnosis or treatment of any clinically symptomatic biochemical or structural abnormality of the GI tract within 6 months prior to screening, or active disease within 6 months prior to screening; including but not limited to cancer, inflammatory bowel disease, diverticulitis, duodenal ulcer, erosive esophagitis, gastric ulcer, pancreatitis (within 12 months of screening), cholelithiasis, amyloidosis, ileus, non-controlled GERD, gastrointestinal obstruction, ischemic colitis or carcinoid syndrome.
* Subject has a history or current evidence of laxative abuse (in the clinical judgment of the physician)
* Hepatic dysfunction (ALT [SGPT] or AST [SGOT] >2.5 times the upper limit of normal) or renal impairment (serum creatinine > 2mg/dL)
* Any evidence of or treatment of malignancy (other than localized basal cell, squamous cell skin cancer or cancer in situ that has been resected) within the previous year
* Any surgery on the stomach, small intestine or colon, excluding appendectomy or cholecystectomy (unless within 60 days of screening visit)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2015-10; Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Rosenbaum, Ph.D., Study Chair — Ardelyx, Inc.
Locations (111):
- United States (111):
  - Ardelyx Investigative Site 149, Birmingham, Alabama
  - Ardelyx Investigative Site 114, Birmingham, Alabama
  - Ardelyx Investigative Site 103, Huntsville, Alabama
  - Ardelyx Investigative Site 100, Huntsville, Alabama
  - Ardelyx Investigative Site 145, Chandler, Arizona
  - Ardelyx Investigative Site 210, Phoenix, Arizona
  - Ardelyx Investigative Site 296, Phoenix, Arizona
  - Ardelyx Investigative Site 277, Tempe, Arizona
  - Ardelyx Investigative Site 269, Tucson, Arizona
  - Ardelyx Investigative Site 187, Tucson, Arizona
  - Ardelyx Investigative Site 199, Tucson, Arizona
  - Ardelyx Investigative Site 140, Harrisburg, Arkansas
  - Ardelyx Investigative Site 274, Little Rock, Arkansas
  - Ardelyx Investigative Site 161, Little Rock, Arkansas
  - Ardelyx Investigative Site 122, Little Rock, Arkansas
  - Ardelyx Investigative Site 129, North Little Rock, Arkansas
  - Ardelyx Investigative Site 105, Canoga Park, California
  - Ardelyx Investigative Site 143, Chula Vista, California
  - Ardelyx Investigative Site 146, Encino, California
  - Ardelyx Investigative Site 147, Encino, California
  - Ardelyx Investigative Site 107, Lomita, California
  - Ardelyx Investigative Site 112, North Hollywood, California
  - Ardelyx Investigative Site 110, Northridge, California
  - Ardelyx Investigative Site 294, San Diego, California
  - Ardelyx Investigative Site 108, Thousand Oaks, California
  - Ardelyx Investigative Site 178, Cutler Bay, Florida
  - Ardelyx Investigative Site 131, Fort Lauderdale, Florida
  - Ardelyx Investigative Site 136, Hialeah, Florida
  - Ardelyx Investigative Site 130, Hialeah, Florida
  - Ardelyx Investigative Site 287, Homestead, Florida
  - Ardelyx Investigative Site 106, Miami, Florida
  - Ardelyx Investigative Site 127, Miami Lakes, Florida
  - Ardelyx Investigative Site 123, Miami Springs, Florida
  - Ardelyx Investigative Site 126, Pompano Beach, Florida
  - Ardelyx Investigative Site 132, Port Orange, Florida
  - Ardelyx Investigative Site 150, St. Petersburg, Florida
  - Ardelyx Investigative Site 254, West Palm Beach, Florida
  - Ardelyx Investigative Site 234, Athens, Georgia
  - Ardelyx Investigative Site 138, Atlanta, Georgia
  - Ardelyx Investigative Site 148, Atlanta, Georgia
  - Ardelyx Investigative Site 137, Norcross, Georgia
  - Ardelyx Investigative Site 213, Savannah, Georgia
  - Ardelyx Investigative Site 124, Snellville, Georgia
  - Ardelyx Investigative Site 157, Boise, Idaho
  - Ardelyx Investigative Site 102, Blue Island, Illinois
  - Ardelyx Investigative Site 162, Evanston, Illinois
  - Ardelyx Investigative Site 202, Oak Lawn, Illinois
  - Ardelyx Investigative Site 259, Topeka, Kansas
  - Ardelyx Investigative Site 192, Crowley, Louisiana
  - Ardelyx Investigative Site 188, Metairie, Louisiana
  - Ardelyx Investigative Site 177, Monroe, Louisiana
  - Ardelyx Investigative Site 198, Zachary, Louisiana
  - Ardelyx Investigative Site 278, Hagerstown, Maryland
  - Ardelyx Investigative Site 255, Towson, Maryland
  - Ardelyx Investigative Site 135, Boston, Massachusetts
  - Ardelyx Investigative Site 267, Brockton, Massachusetts
  - Ardelyx Investigative Site 119, Caro, Michigan
  - Ardelyx Investigative Site 128, Chesterfield, Michigan
  - Ardelyx Investigative Site 224, Saginaw, Michigan
  - Ardelyx Investigative Site 125, Belton, Missouri
  - Ardelyx Investigative Site 156, Billings, Montana
  - Ardelyx Investigative Site 142, Omaha, Nebraska
  - Ardelyx Investigative Site 275, Las Vegas, Nevada
  - Ardelyx Investigative Site 276, Las Vegas, Nevada
  - Ardelyx Investigative Site 182, Las Vegas, Nevada
  - Ardelyx Investigative Site 175, Vineland, New Jersey
  - Ardelyx Investigative Site 293, Albuquerque, New Mexico
  - Ardelyx Investigative Site 151, Brooklyn, New York
  - Ardelyx Investigative Site 170, Great Neck, New York
  - Ardelyx Investigative Site 225, Hartsdale, New York
  - Ardelyx Investigative Site 206, New Windsor, New York
  - Ardelyx Investigative Site 183, New York, New York
  - Ardelyx Investigative Site 226, Asheville, North Carolina
  - Ardelyx Investigative Site 166, Charlotte, North Carolina
  - Ardelyx Investigative Site 205, Fayetteville, North Carolina
  - Ardelyx Investigative Site 104, Greensboro, North Carolina
  - Ardelyx Investigative Site 174, Kinston, North Carolina
  - Ardelyx Investigative Site 280, Winston-Salem, North Carolina
  - Ardelyx Investigative Site 172, Beavercreek, Ohio
  - Ardelyx Investigative Site 223, Cincinnati, Ohio
  - Ardelyx Investigative Site 201, Cincinnati, Ohio
  - Ardelyx Investigative Site 139, Columbus, Ohio
  - Ardelyx Investigative Site 173, Dayton, Ohio
  - Ardelyx Investigative Site 171, Huber Heights, Ohio
  - Ardelyx Investigative Site 117, Mentor, Ohio
  - Ardelyx Investigative Site 247, Springfield, Ohio
  - Ardelyx Investigative Site 144, Jenkintown, Pennsylvania
  - Ardelyx Investigative Site 289, Mt. Pleasant, South Carolina
  - Ardelyx Investigative Site 184, Myrtle Beach, South Carolina
  - Ardelyx Investigative Site 281, North Charleston, South Carolina
  - Ardelyx Investigative Site 261, Sioux Falls, South Dakota
  - Ardelyx Investigative Site 134, Chattanooga, Tennessee
  - Ardelyx Investigative Site 121, Franklin, Tennessee
  - Ardelyx Investigative Site 189, Hermitage, Tennessee
  - Ardelyx Investigative Site 133, Jackson, Tennessee
  - Ardelyx Investigative Site 109, Knoxville, Tennessee
  - Ardelyx Investigative Site 235, Nashville, Tennessee
  - Ardelyx Investigative Site 164, Corpus Christi, Texas
  - Ardelyx Investigative Site 197, Corsicana, Texas
  - Ardelyx Investigative Site 185, Houston, Texas
  - Ardelyx Investigative Site 120, Houston, Texas
  - Ardelyx Investigative Site 113, McKinney, Texas
  - Ardelyx Investigative Site 111, Plano, Texas
  - Ardelyx Investigative Site 118, Plano, Texas
  - Ardelyx Investigative Site 101, San Antonio, Texas
  - Ardelyx Investigative Site 240, San Antonio, Texas
  - Ardelyx Investigative Site 159, Orem, Utah
  - Ardelyx Investigative Site 207, Sandy City, Utah
  - Ardelyx Investigative Site 155, South Ogden, Utah
  - Ardelyx Investigative Site 231, Norfolk, Virginia
  - Ardelyx Investigative Site 141, Richmond, Virginia

REFERENCES:
- [Derived] Lacy BE, Shin AS, Cangemi DJ, Yang Y, Zhao S, Rosenbaum DP. Tenapanor is associated with earlier and sustained symptom relief in IBS-C: a post hoc analysis. Therap Adv Gastroenterol. 2026 Jan 24;19:17562848251414831. doi: 10.1177/17562848251414831. eCollection 2026. PMID 41601848
- [Derived] Lembo AJ, Friedenberg KA, Fogel RP, Edelstein S, Zhao S, Yang Y, Rosenbaum DP, Chey WD. Long-term safety of tenapanor in patients with irritable bowel syndrome with constipation in the T3MPO-3 study. Neurogastroenterol Motil. 2023 Nov;35(11):e14658. doi: 10.1111/nmo.14658. Epub 2023 Sep 5. PMID 37668173
- [Derived] Chey WD, Lembo AJ, Yang Y, Rosenbaum DP. Efficacy of Tenapanor in Treating Patients With Irritable Bowel Syndrome With Constipation: A 26-Week, Placebo-Controlled Phase 3 Trial (T3MPO-2). Am J Gastroenterol. 2021 Jun 1;116(6):1294-1303. doi: 10.14309/ajg.0000000000001056. PMID 33337659
- [Derived] Chey WD, Lembo AJ, Rosenbaum DP. Efficacy of Tenapanor in Treating Patients With Irritable Bowel Syndrome With Constipation: A 12-Week, Placebo-Controlled Phase 3 Trial (T3MPO-1). Am J Gastroenterol. 2020 Feb;115(2):281-293. doi: 10.14309/ajg.0000000000000516. PMID 31934897

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period
Arm/Group | 50mg BID | Placebo
Started | 307 | 299
Completed | 261 | 272
Not Completed | 46 | 27
Period: Randomized Withdrawal Period
Arm/Group | 50mg BID | Placebo
Started | 261 | 272
Completed | 250 | 260
Not Completed | 11 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 50mg BID | Placebo | Total
Number analyzed (Participants) | 307 | 299 | 606
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (13.38) | 44.9 (13.04) | 45 (13.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 244 | 249 | 493
  Male | 63 | 50 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 98 | 83 | 181
  Not Hispanic or Latino | 209 | 216 | 425
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 10 | 4 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 88 | 100 | 188
  White | 201 | 186 | 387
  More than one race | 8 | 7 | 15
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.88 (7.198) | 29.30 (6.442) | 29.60 (6.836)

OUTCOME MEASURES:

1. Primary Outcome: 6 of 12 Week Overall Responder Rate
Description: An overall responder is defined as a weekly responder for the first 6/12 weeks where both CSBM and abdominal pain response criteria were met for the week. The CSBM response criteria are defined as an increase of one or more change in average weekly CSBMs from baseline. The definition of a CSBM is as follows: A CSBM is a spontaneous bowel movement (SBM) for which the subject responds "yes" to the following question; "Did you feel like you completely emptied your bowels?" The abdominal pain response criterion is defined as a decrease of 30% or more of percent change in average weekly worst abdominal pain from baseline.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg BID | Placebo
Number analyzed (Participants) | 307 | 299
Participants | 83 | 56
Statistical Analysis 1: Comparison: 50mg BID vs Placebo; Test type: Superiority; p < 0.02, Cochran-Mantel-Haenszel; Risk Difference (RD) = 8.31

2. Secondary Outcome: 6 of 12 Week Overall Complete Spontaneous Bowel Movement (CSBM)Responder Rate
Description: An overall CSBM responder is defined as a weekly responder for the first 6/12 weeks. The CSBM response criteria are defined as an increase of one or more change in average weekly CSBMs from baseline. The definition of a CSBM is as follows: A CSBM is a spontaneous bowel movement (SBM) for which the subject responds "yes" to the following question; "Did you feel like you completely emptied your bowels?"
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg BID | Placebo
Number analyzed (Participants) | 307 | 299
Participants | 104 | 88

3. Secondary Outcome: 6 of 12 Week Overall Abdominal Pain Responder Rate
Description: An overall abdominal pain responder is defined as a weekly responder for the first 6/12. The abdominal pain response criterion is defined as a decrease of 30% or more of percent change in average weekly worst abdominal pain from baseline.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg BID | Placebo
Number analyzed (Participants) | 307 | 299
Participants | 135 | 99
Statistical Analysis 1: Comparison: 50mg BID vs Placebo; Test type: Superiority; p < 0.008, Cochran-Mantel-Haenszel; Risk Difference (RD) = 10.86

4. Secondary Outcome: 9 of 12 Week Overall Responder Rate
Description: An overall responder is defined as a weekly responder for the first 9/12 weeks where both CSBM and abdominal pain response criteria were met for the week. The CSBM response criteria are defined as an increase of one or more change in average weekly CSBMs from baseline and a minimum of at least 3 CSBMs that same week. The definition of a CSBM is as follows: A CSBM is a spontaneous bowel movement (SBM) for which the subject responds "yes" to the following question; "Did you feel like you completely emptied your bowels?" The abdominal pain response criterion is defined as a decrease of 30% or more of percent change in average weekly worst abdominal pain from baseline.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg BID | Placebo
Number analyzed (Participants) | 307 | 299
Participants | 42 | 10
Statistical Analysis 1: Comparison: 50mg BID vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 10.34

5. Secondary Outcome: 9 of 12 Week Overall CSBM Responder Rate
Description: An overall CSBM responder is defined as a weekly responder for the first 9/12 weeks. The CSBM response criteria are defined as an increase of one or more change in average weekly CSBMs from baseline and a minimum of at least 3 CSBMs that same week. The definition of a CSBM is as follows: A CSBM is a spontaneous bowel movement (SBM) for which the subject responds "yes" to the following question; "Did you feel like you completely emptied your bowels?"
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg BID | Placebo
Number analyzed (Participants) | 307 | 299
Participants | 52 | 15
Statistical Analysis 1: Comparison: 50mg BID vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 11.92

6. Secondary Outcome: 9 of 12 Week Overall Abdominal Pain Responder Rate
Description: An overall abdominal pain responder is defined as a weekly responder for the first 9/12 weeks. The abdominal pain response criterion is defined as a decrease of 30% or more of percent change in average weekly worst abdominal pain from baseline.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg BID | Placebo
Number analyzed (Participants) | 307 | 299
Participants | 93 | 58
Statistical Analysis 1: Comparison: 50mg BID; Test type: Superiority; p < 0.003, Cochran-Mantel-Haenszel; Risk Difference (RD) = 10.9

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | 50mg BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/307 | 0/299
Serious Adverse Events (participants affected / at risk) | 6/307 | 0/299
Other Adverse Events (participants affected / at risk) | 45/307 | 5/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50mg BID (N=307) | Placebo (N=299)
Panick Attack (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol withdrawal syndromw (Psychiatric disorders) | 1 (1) | 0 (0)
Major Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pineal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50mg BID (N=307) | Placebo (N=299)
Diarrhea (Gastrointestinal disorders) | 45 (45) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-08-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT02621892/Prot_000.pdf
  • Statistical Analysis Plan (2015-12-16): https://cdn.clinicaltrials.gov/large-docs/92/NCT02621892/SAP_001.pdf